CLINICAL TRIAL: NCT05354193
Title: Analysis of microRNAs Expression in Patients Who Evolved to Vasoplegic Syndrome After On-pump Coronary Artery Bypass Surgery
Brief Title: Analysis of miRNAs Expression in Vasoplegic Syndrome After On-pump Coronary Artery Bypass Surgery
Acronym: PREVENT
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); InCor Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 4435/16/101
Record Dates: First submitted 2018-01-10; First posted 2022-04-29 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2018-01

CONDITIONS: Vasoplegic Syndrome; Vasoplegia; Surgery-Complications; Surgery; Cardiovascular Diseases; Cardiovascular Morbidity
Keywords: vasoplegic syndrome; vasoplegic; surgery; cardiovascular; microRNAs; miRNAs
MeSH Terms: conditions — Vasoplegia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 3 milliliters of venous blood will be collected before CPB, 3 milliliters of venous blood 15 minutes after the reversal of heparin with protamine and a small fragment of aortic tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vasoplegic syndrome: Patients undergoing on-pump coronary artery bypass graft who develops vasoplegic syndrome 24 - 48 hours after surgery.
  Interventions: Other: vasoplegic syndrome
- control: Patients undergoing on-pump coronary artery bypass graft who does not develop vasoplegic syndrome.
  Interventions: Other: vasoplegic syndrome

INTERVENTIONS:
Other: vasoplegic syndrome — In all included patients, 3 milliliters of venous blood will be collected before cardiopulmonary bypass, 3 milliliters of venous blood 15 minutes after the reversal of heparin with protamine and a small fragment of aortic tissue. Samples of biological material will be compared between the control and vasoplegic groups for the difference in amount and type of miRNA present.
  For the diagnosis of vasospastic syndrome, the following criteria were adopted: mean arterial pressure < 65 mmHg, cardiac index < 2.2 L / min / m2, refractory to replacement of at least 1000 milliliters of crystalloid, excluding other causes such as tamponade, bleeding and cardiogenic shock

SUMMARY:
This study looks for a correlation between microRNAs (miRNAs) and vasoplegic syndrome after on-pump coronary artery bypass surgery.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are among the main causes of morbidity and mortality in the world, and in Brazil they account for approximately 31% of all causes of death and 42% of deaths due to noncommunicable diseases. In 2014 were carried out a total number of 92,000 heart surgeries in Brazil and these are usually performed using Cardiopulmonary Bypass (CPB), which is made by the diversion of blood circulation of the lungs and heart to a heart-lung machine, which keeps cardio circulatory functions and oxygenates the blood. Despite enable various types of major cardiac surgery, the use of CPB can cause serious side effects such as post perfusion vasoplegic syndrome (VS). This is characterized by increased cardiac output, hypotension, systemic inflammatory response and decreased vascular resistance, affecting 9-44% of patients in the postoperative period of cardiac surgery, with a mortality of 27%. Treatment to VS are limited and the drugs are often ineffective, including noradrenaline, vasopressin, and methylene blue. Another difficulty encountered by the surgeon is to establish a predictive factor for VS. Systems risk predictors that use score and are well validated as EuroSCORE (European System for Cardiac Operative Risk Evaluation) have not been tested for VS. Much has been studied on the use of biomarkers as predictors and for prognosis as well as to improve predictive power of the rating systems available. MicroRNAs (miRNAs) are noncoding RNA molecules that control gene expression in the intracellular environment and are present circulating in various body fluids including peripheral blood. These molecules can be used as biomarkers of various pathologies including CVD. Despite the existence of numerous studies that demonstrate the importance of miRNAs in the development of CVDs. There are no studies that address the issue in VS. Therefore, the objective of the project is to identify the presence of blood miRNAs that are altered in patients with pre and intra-operative cardiovascular surgery and assess whether these miRNAs can be used as predictors and biomarkers of mortality for VS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who go to coronary artery by-pass , on-pump surgery
* Patients who sign an informed consent
* Only elective or urgency surgery

Exclusion Criteria:

* off-pump surgery
* emergency surgery
* previous use of vasoactive drugs or Intra aortic balloon
* Patients with active acute coronary syndrome
* Acute mesenteric ischemia, Reynaud disease, neoplasia and Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our population is build whith both sexy, bigger than 18 years old, who has indication of coronary artery surgery. that was selected.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Profile of miRNA | 6 months
  Find out if it is possible to use mirna as a predictor of vasoplegic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Omar Mejía, Principal Investigator — InCor Heart Institute; Renato Cesar de Souza, Principal Investigator — InCor Heart Institute; Edecio Cunha-Neto, Principal Investigator — InCor Heart Institute; Fábio Jatene, Study Chair — InCor Heart Institute; Ludmila Ferreira, Principal Investigator — Federal University of Minas Gerais; Bianca Meneguini, Principal Investigator — InCor Heart Institute
Locations (1):
- Omar Asdrubal Vilca Mejia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided